CLINICAL TRIAL: NCT06297694
Title: Clinical Interpretation and Cutoff Scores for Manual Ability Measured by the ABILHAND Questionnaire in Individuals With Rheumatoid Arthritis
Brief Title: Clinical Interpretation and Cutoff Scores for ABILHAND Questionnaire in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Berna Cagla Balkisli, Principal Investigator, Pamukkale University
Other Study IDs: PamukkaleU.
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In individuals with rheumatoid arthritis, the most significant symptom is the loss of manual ability and function in the hands. In rheumatoid arthritis, where patient-reported assessment scales are frequently used, hand skills should be evaluated with an ideal questionnaire that best represents hand activities. The ABILHAND-RA questionnaire possesses all these features, being a short and easily fillable survey. The aim is to determine of clinically significant cutoff scores for perceived manual ability evaluated by ABILHAND corresponding to observed and perceived upper extremity assessments in individuals with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* People between the ages of 20-65, who were diagnosed with RA according to ACR criteria by the PAU Rheumatology clinic and who volunteered to participate in the study, will be included.

Exclusion Criteria:

* Patients with RA who have a neurological disease that may affect hand functions (peripheral nerve lesion, trauma, operation, cerebrovascular accident), a psychiatric disease that affects cooperation, heart failure and lung pathology that affect daily living activities, and those with other concurrent autoimmune and rheumatic diseases.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAU Romatology clinic
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score (DAS 28) | Baseline
  It is used to evaluate disease activity in individuals with rheumatoid arthritis. DAS28 is a tool consisting of 28 tender joint count (range 0-28), 28 swollen joint count (range 0-28), ESR (erythrocyte sedimentation rate) and overall health assessment on a visual analogue scale (range 0-100). The level of disease activity is low It is interpreted as (DAS28 ≤3.2), medium (3.2< DAS28 ≤ 5.1) or high (DAS28 > 5.1).
Nine hole peg test | Baseline
  It is a battery that aims to measure the loss of skills in the hand. This device is a device consisting of a square platform and a storage box. There are 9 holes in the square area (12.7x2cm) and 9 cylinders suitable for these holes. The diameter of the holes was 0.71 cm, the diameter of the cylinders was 0.64 cm, the length was 3.2 cm, the distance between the holes was 3.2 cm, the hole depth was 1.3 cm and the size of the storage box was 13x13 cm. What is requested from the patients is to quickly take the 9 cylinders from the storage box, place them in the holes, quickly remove them from the holes and place them in the storage box, without taking a break. Meanwhile, the time is measured in seconds with a stopwatch. Three separate measurements will be made for the right and left hand and the average will be taken.
Hand grip strength | Baseline
  Grip strength in the dominant and non-dominant hand will be evaluated in 'kg' unit with a JAMAR (Sammons Preston, USA) hand dynamometer. Patients will be measured in a sitting position with the elbow flexed at 90° and the wrist in the mid-position with the thumb pointing up. The measurement will be made three times consecutively and the average value will be used. Values will be recorded in kilogram units.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Basakci Calik, Study Director — Pamukkale University
Locations (1):
- Pamukkale University School of Physical Therapy and Rehabilitation, Denizli, Turkey (Türkiye)